CLINICAL TRIAL: NCT00823784
Title: Prospective Randomized Trial Comparing Transanal Doppler de-Arterialization (THD) Versus Stapler Operation for 3rd Degree Hemorrhoids
Brief Title: Prospective Randomized Trial Comparing THD Versus Stapler Operation for 3rd Degree Hemorrhoids
Acronym: THD/stapler
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Societa Italiana di Chirurgia ColoRettale (Network)
Responsible Party: Aldo Infantino, Societa Italiana di Chirurgia ColoRettale
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Siccr trial THD/stapler
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Hemorrhoids
Keywords: hemorrhoids; stapler; Doppler; artery ligation; outcome; recurrence
MeSH Terms: conditions — Hemorrhoids; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1THD group (Experimental): Series of 135 patients with 3rd degree Hemorrhoids treated by THD device under spinal anaesthesia
  Interventions: Procedure: Transanal doppler hemorrhoidal ligation
- 2 stapler group (Active Comparator): 135 patients with 3rd degree hemorrhoids will be treated by staple hemorrhoidopexy
  Interventions: Procedure: stapled hemorrhoidopexy

INTERVENTIONS:
Procedure: Transanal doppler hemorrhoidal ligation — THD technique involves identification and ligation of the terminal hemorrhoid arteries (about 6) followed by mucopexy
  Other Names: THD technique
  Arms: 1THD group
Procedure: stapled hemorrhoidopexy — Staple hemorrhoidopexy involves resection of a ring of low rectal mucosa an lifting the hemorrhoids up in the anal canal with a stapled suture
  Other Names: Longo's technique
  Arms: 2 stapler group

SUMMARY:
Haemorrhoids have, in literature, extremely high ranges of prevalence, 4,4% to 36% and there is a debate on the best treatment for III degree hemorrhoids. The Stapled Hemorrhoidopexy is indicated in grade III haemorrhoids due to its advantages vs. other techniques in pain reduction and time before resume of normal activity. The new technique of Doppler guided trans-anal arterial ligation (THD) appear to be another important therapeutic tool thanks to its scarce complications, the minimally invasive procedure and efficacy of the short term results. The rationale of the two surgical techniques is different: in fact, the Stapled Hemorrhoidopexy is based on the hypothesis that the mucosal and sub/mucosal resection and stapling can cure the prolapse, etiologic factor of haemorrhoids; on the other hand, the interruption of the arterial inflow of hemorrhoids by THD reduces hemorrhoidal tissue." Aim of this study is to compare 2 techniques: The doppler guided transanal haemorrhoidal dearterialisation with the THD device and the stapled Haemorrhoidopexy (according to Longo) for III degree (Goligher) haemorrhoid, not regarding the number of prolapsed piles

DETAILED DESCRIPTION:
After informed consent 284 patients with III degree hemorrhoids from 10 colorectal units will be randomized into two groups: stapler vs doppler guided transanal hemorrhoidal dearterialisation with the THD device.The early and long term outcome, as well as other secondary outcomes (costs, return to work and degree of satisfaction) will be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* III degree hemorrhoids
* both sex
* age between 18 and 70 years
* ability to understand the procedure
* written informed consent

Exclusion Criteria:

* previous surgery for hemorrhoids
* fecal incontinence
* obstructed defecation
* other active anorectic diseases
* irritable bowel syndrome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2008-01; Primary Completion 2009-01 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
early complication rate (bleeding, pain) and long term outcome (symptomatic hemorrhoids recurrence) after stapled hemorrhoidopexy versus transanal hemorrhoid arteries ligation and mucopexy | early postoperative period (30 days) and after 1 year

SECONDARY OUTCOMES:
Time to return to the working activities, costs for the public health system and the degree of patients' satisfaction | early postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Donato F Altomare, MD, Study Chair — Societa Italiana di Chirurgia ColoRettale
Locations (1):
- Santa Maria dei Battuti Hospital, S Vito Al Tagliamento, PN, Italy

REFERENCES:
- [Background] Dal Monte PP, Tagariello C, Sarago M, Giordano P, Shafi A, Cudazzo E, Franzini M. Transanal haemorrhoidal dearterialisation: nonexcisional surgery for the treatment of haemorrhoidal disease. Tech Coloproctol. 2007 Dec;11(4):333-8; discussion 338-9. doi: 10.1007/s10151-007-0376-4. Epub 2007 Dec 3. PMID 18060529